CLINICAL TRIAL: NCT00692107
Title: Phase III Study for Prostate Cancer, Randomizing Between Two Radiation Dose Levels (68 Gy vs. 78 Gy) and Utilizing Three Dimensional Conformal Radiotherapy
Brief Title: Radiotherapy for Prostate Cancer: Conventional Dose Versus High Dose
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Erasmus Medical Center (Other); Dutch Cancer Society (Other)
Responsible Party: Dr. J. Lebesque, Dr. P. Koper, Erasmus Medical Center / The Netherlands Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CKVO 96-10
Record Dates: First submitted 2005-08-25; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Prostatic Neoplasms
Keywords: Radiotherapy; Dose
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiation Dosage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 68 Gy
  Interventions: Radiation: Gray
- 2 (Experimental): 78 Gy
  Interventions: Radiation: Gray

INTERVENTIONS:
Radiation: Gray — 68 Gy vs. 78 Gy
  Arms: 1
Radiation: Gray — 68 Gy vs. 78 Gy
  Arms: 2

SUMMARY:
3-D conformal radiotherapy offers the opportunity to reach higher tumor doses with acceptable complication rates compared to conventional radiotherapy. There are retrospective and preliminary prospective reports of a better local control / disease free survival (including PSA control) using higher tumor doses. A prospective randomised phase III study is required to validate these reports. The purpose of this randomized phase III study is to investigate and compare the tumor control and toxicity in prostate cancer patients treated to 68 Gy and 78 Gy;

DETAILED DESCRIPTION:
Patients were stratified by hospital, treatment group, age and (neo)adjuvant hormonal therapy. Four treatment groups with specific radiation volumes were defined depending on the estimated risk of tumour involvement of the seminal vesicles (based on T-stage, initial PSA and Gleason Score or Differentiation Grade).The dose was delivered with daily fractions of 2 Gy, five times a week. The total duration of the treatment was 7 weeks for patients treated to 68 Gy and 8 week for 78 Gy.

Objectives:

* To test in a phase III randomised study the hypothesis that higher radiation doses lead to a higher freedom from failure rate for localized prostate cancer.
* To test the hypothesis that a higher freedom from failure rate leads to a longer disease-free survival and overall survival.
* To limit acute and late toxicity with respect to gastro-intestinal and urological toxicity.
* To evaluate different PSA related endpoints for local failure and distant metastasis.
* To establish a database of patients treated to escalated doses with Dose Volume Histograms of the normal tissues at risk for each individual patient and common toxicity endpoints.
* To validate a model to estimate normal tissue complication probabilities (NTCPs) of rectum and bladder, based on the above-mentioned database, and to obtain reliable parameter values for NTCP estimations.

ELIGIBILITY:
Inclusion Criteria:

* locally confined adenocarcinoma of the prostate
* all T-stages with a PSA < 60ng/ml, except any T1a tumor and well-differentiated (or Gleason score < 5) T1b-c tumors with PSA-levels ≤ 4 ng/ml
* Karnofsky Performance Status of 80 or more

Exclusion Criteria:

* distant metastases
* positive regional lymph nodes proven by surgical or cytological sampling
* on anticoagulants
* previous prostatectomy
* previous pelvic irradiation

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 1997-06; Primary Completion 2005-05 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Freedom from failure

SECONDARY OUTCOMES:
Toxicity
Overall survival
Freedom from clinical failure

CONTACTS AND LOCATIONS:
Overall Officials: Joos V Lebesque, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (4):
- Netherlands (4):
  - The Netherlands Cancer Institute, Amsterdam
  - Zeeuws Radiotherapeutic Institute, Flushing
  - Radiotherapeutic Institute Friesland, Leeuwarden
  - Daniel Den Hoed Cancer Center, Rotterdam

REFERENCES:
- [Result] Peeters ST, Heemsbergen WD, van Putten WL, Slot A, Tabak H, Mens JW, Lebesque JV, Koper PC. Acute and late complications after radiotherapy for prostate cancer: results of a multicenter randomized trial comparing 68 Gy to 78 Gy. Int J Radiat Oncol Biol Phys. 2005 Mar 15;61(4):1019-34. doi: 10.1016/j.ijrobp.2004.07.715. PMID 15752881
- [Result] Peeters ST, Hoogeman MS, Heemsbergen WD, Slot A, Tabak H, Koper PC, Lebesque JV. Volume and hormonal effects for acute side effects of rectum and bladder during conformal radiotherapy for prostate cancer. Int J Radiat Oncol Biol Phys. 2005 Nov 15;63(4):1142-52. doi: 10.1016/j.ijrobp.2005.03.060. Epub 2005 Jun 4. PMID 15939547
- [Derived] Kim S, Kong JH, Lee Y, Lee JY, Kang TW, Kong TH, Kim MH, You SH. Dose-escalated radiotherapy for clinically localized and locally advanced prostate cancer. Cochrane Database Syst Rev. 2023 Mar 8;3(3):CD012817. doi: 10.1002/14651858.CD012817.pub2. PMID 36884035
- [Derived] Heemsbergen WD, Al-Mamgani A, Slot A, Dielwart MF, Lebesque JV. Long-term results of the Dutch randomized prostate cancer trial: impact of dose-escalation on local, biochemical, clinical failure, and survival. Radiother Oncol. 2014 Jan;110(1):104-9. doi: 10.1016/j.radonc.2013.09.026. Epub 2013 Nov 15. PMID 24246414